CLINICAL TRIAL: NCT06999577
Title: The MVP Trial: A Randomized Controlled Trial of Mechanism Guided vs PPI Strategy for Laryngopharyngeal Reflux
Brief Title: The Mechanism Versus PPI Trial
Acronym: MVP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rena Yadlapati, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 807412; R01DK139089 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Laryngopharyngeal Reflux; Cough; Throat Clearing; Dysphonia; Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux; Cough; Dysphonia; Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: 8 week intervention with a daily oral capsule (omeprazole 40mg or placebo) and 3 intervention visits at week 1, 4, and 8.
Who Masked: Participant, Care Provider
Masking Description: The participant will not know which strategy group they are randomized to and they will not know which daily oral capsule (omeprazole 40mg or placebo) they have been dispensed. The study provider they meet with during intervention visits will not know the results of their upper endoscopy and reflux testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mechanism Guided Strategy (Active Comparator): 1) 8-week course of double dose PPI or placebo; 2) Laryngeal Recalibration Therapy (LRT) with speech language pathologist (SLP). Subjects will receive PPI if their reflux monitoring is consistent with GERD and placebo if it is not consistent with GERD. SLP will administer LRT: LRT utilizes therapies that SLPs standardly utilize (mechanical and cognitive guidance) in combination specifically designed to treat laryngeal symptoms.
  1. Mechanical Guidance: The SLP will guide subjects through laryngeal suppression, changing voice production, and improving breath coordination.
  2. Cognitive Guidance: The SLP will guide subjects through relaxation and conceptualization changes.
  3. Lifestyle Recommendations: In addition to receiving LRT, subjects will be counseled on typical lifestyle recommendations for GERD, detailed in the Usual Care Strategy below.
  Interventions: Drug: Omeprazole 40 MG; Behavioral: Laryngeal Recalibration Therapy; Behavioral: GERD Lifestyle Recommendations
- Usual Care Strategy (Active Comparator): 1) an 8-week course of double dose PPI and 2) lifestyle counseling. This represents the control group receiving usual care and will serve as the study's active control group. In order to maintain group concealment, subjects will receive counseling from a study investigator on standard lifestyle modifications recommended for GERD at intervals mirroring that of the mechanism guided strategy: week 1, week 4, and week 8 which is also reflective of standard recommended follow-up and counseling in GERD management.
  Interventions: Drug: Omeprazole 40 MG; Behavioral: GERD Lifestyle Recommendations

INTERVENTIONS:
Drug: Omeprazole 40 MG — 8 week double dose therapy of proton pump inhibitor or placebo.
  Other Names: Prilosec; NDA 21-229
Behavioral: Laryngeal Recalibration Therapy — LRT utilizes therapies that SLPs standardly utilize (mechanical and cognitive guidance) in combination specifically designed to treat laryngeal symptoms. Each session with the SLP will guide subjects through these therapies. The existing script-based LRT protocol consists of the following: 1) mechanical guidance (laryngeal suppression, voice production, breath coordination), 2) cognitive guidance (identification of thinking patterns, recalibration of thoughts about laryngeal sensations).
  Other Names: LRT
  Arms: Mechanism Guided Strategy
Behavioral: GERD Lifestyle Recommendations — This is the typical lifestyle recommendations for GERD used clinically.

SUMMARY:
The goal of this clinical trial is to learn if a mechanism guided strategy that utilizes a multidisciplinary approach to treat adults patients (age 18-89) with chronic throat symptoms who are undergoing clinical evaluation for laryngopharyngeal reflux (LPR) is more effective than the usual care strategy with proton pump inhibitor (PPI) therapy used in gastroenterology for these patients.

The main question it aims to answer is: Will a greater proportion of the mechanism guided strategy participants achieve symptom response in comparison to the usual care strategy participants?

If there is a comparison group: Researchers will compare the mechanism guided strategy to usual care strategy to see if treatment response differs between the groups.

Participants will be be asked to do the following:

* participate in an 8-week blinded study phase where they will be randomized to either 1) Mechanism Guided Strategy or 2) Usual Care Strategy
* take an oral capsule daily (omeprazole 40mg or placebo)
* come to 3 in-person visits at UC San Diego Health for an intervention visit with a study provider
* consider incorporating recommended lifestyle modifications
* complete weekly surveys

DETAILED DESCRIPTION:
This research study is being conducted to compare the efficacy between usual care and a novel mechanism guided strategy for adults with chronic throat (laryngeal) symptoms undergoing evaluation for laryngopharyngeal reflux (LPR).

Usual care strategy is used clinically and is known to reduce chronic throat symptoms. The mechanism guided strategy is a new treatment that personalizes the application of acid suppression medication and voice therapy to the patient. The mechanism guided strategy is being evaluated for how well it works in patients with these throat symptoms.

Participants who are undergoing clinical evaluation for laryngopharyngeal reflux (LPR) inclusive of an upper endoscopy with ambulatory pH monitoring (reflux testing) will be recruited for participation in this study.

Participants will undergo screening to confirm eligibility. Once informed consent is administered and signed, participants will be asked about their demographic background, current symptoms, brief medical history, and current medications. Screening takes place within 30 days of a participant's scheduled clinical upper endoscopy with reflux testing.

After completing the clinical upper endoscopy and reflux testing, they will be scheduled for their first intervention visit, about 1 week later.

Participants will be randomized to 1 of 2 arms with of the study: 1) Mechanism Guided Strategy or 2) Usual Care Strategy. Randomization is 1:1 based on permuted block randomization in REDCap to mechanism guided or usual care strategy with stratification by concomitant esophageal + laryngeal symptoms versus isolated laryngeal symptoms.

Participants will then attend 3 in person treatment visits at UC San Diego Health's Research Clinic.

Participants will undergo measures at these visits included: 1) acoustics, 2) aerodynamics, 3) patient reported outcomes measuring symptom burden and quality of life, 4) Fasting saliva samples for pepsin and bile acid analysis, and 5) physiologic measures. The study team will also collect height, weight, current medications, and adverse events. Participants will be dispensed an oral capsule (omeprazole 40mg or placebo) based on their randomly assigned strategy. The participants in the mechanism guided strategy will receive omeprazole 40mg daily if their clinical upper endoscopy and reflux testing are conclusive with GERD. They will receive placebo if their upper endoscopy and reflux testing are not conclusive with GERD. The participants in the usual care strategy will receive omeprazole 40mg daily regardless of the results of their upper endoscopy and reflux testing.

Participants will meet with a study provider who will administer treatment according to assigned arm and provide recommended lifestyle modifications.

Participants will complete an online survey weekly to indicate if they have taken their oral capsule daily and if they have incorporated recommended lifestyle modifications.

Intervention visits will take place during week 1, week 4, and week 8. After the week 8 intervention visit is complete, participants will be told which strategy they were assigned to, if they are taking omeprazole 40mg or placebo, and be transitioned back to clinical care.

The most common risks or discomforts of this study are emotional upset during symptom reflection and side effects of omeprazole. The most serious risks include side effects of omeprazole which include generally mild side effects: headache, abdominal pain, nausea, diarrhea, vomiting, and flatulence.

ELIGIBILITY:
Inclusion Criteria:

1. 18-89 years of age
2. >8 weeks of laryngeal symptoms (cough, throat clearing, dysphonia)
3. Standard evaluation for LPR, undergoing EGD (with endoscopic evaluation of the hypopharynx) and reflux monitoring off acid suppression
4. Off acid suppression therapy for at least 2 weeks prior to randomization.

Exclusion Criteria:

1. PPI intolerance and/or known hypersensitivity to the formulation or substituted benzimidazoles
2. History of foregut surgery
3. Known diagnosis of achalasia
4. Inability to fast for 4 hours (no food or drink)
5. Active tobacco use
6. Pregnant or breastfeeding
7. Unable to consent in English or Spanish
8. Unable to provide consent without a legal guardian or representative
9. Imprisoned
10. Endoscopic findings conclusive with esophageal mucosal abnormalities
11. Unable to proceed with reflux monitoring
12. Use of acid suppression during the reflux monitoring and/or before the study medication (omeprazole or placebo) is dispensed
13. Prior LRT for reflux related symptoms
14. History of major psychiatric comorbidity
15. Unable to attend in person study visits at UCSD

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Response | 5 years
  Proportion of subjects with symptom response measured by the reflux symptom index (RSI) score.

SECONDARY OUTCOMES:
Diagnostic Methods for LPR | 5 years
  Symptom response to PPI measured by the RSI score

CONTACTS AND LOCATIONS:
Overall Officials: Rena Yadlapati, MD, Principal Investigator — UC San Diego Health
Locations (1):
- University of California San Diego, San Deigo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
This study has a data management and sharing plan. The study data will be submitted to a generalist repository that is participating in the NIH Generalist Repository Ecosystem Initiative.
Supporting Information: Study Protocol, CSR
Time Frame: The dataset will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: To maximize the appropriate sharing of scientific data and protect research participants' privacy and confidentiality, reuse of this dataset should use the following Data Use Limitations (DULs) under Controlled Access that is made available by a data repository only after approval of the request by the UCSD Health review panel process.
  * Health/Medical/Biomedical - The dataset can only be used for studying health, medical, or biomedical conditions and does not include the study of population origins or ancestry.
  * IRB Approval Required (IRB) - The requesting institution's IRB or equivalent body must approve the requested use.